CLINICAL TRIAL: NCT04242771
Title: Neurophysiological Patterns of Mindfulness Meditation for Insomnia
Brief Title: Mindfulness Meditation for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P000984
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants will utilize a daily sleep program available within a widely used smartphone app, which includes seven soundtracks (10-15min each) for guided mindfulness practice at bedtime. Techniques include breathing exercises, mental imagery, awareness of body and mind, and muscle and body relaxation.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Subjects practice mindfulness before bedtime

SUMMARY:
This is a pilot study evaluating the feasibility and acceptability of a non-pharmacological, mind-body intervention to improve sleep quality, including a preliminary evaluation of neurophysiological signals. The study involves 4 weeks of guided mind-body practice at home using a smartphone app during bedtime and pre/post in-lab sleep study visits.

ELIGIBILITY:
Inclusion Criteria:

* 1. age 20 - 50 years*
* 2. chronic insomnia (defined by Diagnostic and Statistical Manual Diploma in Social Medicine, DSM-V or International Classification of Sleep Disorders - Third Edition, ICSD-3) with sleep latency >20 minutes
* 3. speak and understand English
* 4. have a smart phone for mobile app installation

Exclusion Criteria:

* 1. sleep disorders other than insomnia (e.g., narcolepsy, restless leg syndrome, sleep deprivation, jet lag, etc)
* 2. shift worker or routine night shifts
* 3. women with pregnancy or breast feeding
* 4. history of head trauma or surgery
* 5. regular (defined as twice a week or more) practice of mind-body interventions
* 6. neurological disorders (e.g. epilepsy, dementia, stroke, Parkinson's disease, neuroinfections, brain tumors, etc.)
* 7. current use of neurologic, psychiatric, or cardiovascular medications that have expected neuropsychiatric or cardiovascular effects (i.e., beta-blockers, hypnotics, antidepressants).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (i.e., subject retention at initial follow-up assessment) | At one month follow up visit
  The primary metric for assessing Feasibility will be subject retention at the initial follow-up assessment. This includes the proportion of enrolled subjects that are active in the study at the initial follow-up assessment.

SECONDARY OUTCOMES:
Acceptability | At completion of the 4 week program
  The primary metric for assessing Acceptability will be a self-report Acceptability questionnaire which evaluates enjoyableness, convenience, helpfulness, relevancy, odds of future use, and overall satisfaction of the program.

OTHER OUTCOMES:
Insomnia Severity Index | At baseline and at the end of 4-week program
  A commonly used subjective sleep measure
Polysomnogram-derived sleep onset latency | At baseline and at the end of 4-week program
  The amount of time it takes to fall asleep after the lights have been turned off.
Polysomnogram-derived sleep efficiency | At baseline and at the end of 4-week program
  Sleep efficiency is the ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No